CLINICAL TRIAL: NCT03416829
Title: Preliminary Study 1 to Test the Effects of Ambulatory Voice Biofeedback in Small Groups of Patients With Vocal Hyperfunction
Brief Title: Preliminary Study 1 to Test the Effects of Ambulatory Voice Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Robert E Hillman, Research Director at the MGH Voice Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002849A; 1P50DC015446-01A1 (NIH)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Vocal Fold Nodules
Keywords: Ambulatory; Biofeedback; Voice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100% frequency (Experimental): Some patients will be assigned (via block randomization) to receive ambulatory voice biofeedback (100% frequency - vibrotactile cueing every time the participant exceeds a vocal intensity threshold). Voice monitoring will be conducted for 3 days (device automatically turns off after 42 minutes of voicing): Day 1: biofeedback will be active all day , Day 2: the day after Day 1, no biofeedback, just monitoring to test short-term retention. Day 3: 7 days post-Day 1, no biofeedback, just monitoring to test longer-term retention.
  Interventions: Behavioral: Ambulatory voice biofeedback
- 25% frequency (Experimental): Some patients will be assigned (via block randomization) to receive ambulatory voice biofeedback (25% frequency - vibrotactile cueing every 4th time the participant exceeds a vocal intensity threshold). Voice monitoring will be conducted for 3 days (device automatically turns off after 42 minutes of voicing): Day 1: biofeedback will be active all day , Day 2: the day after Day 1, no biofeedback, just monitoring to test short-term retention. Day 3: 7 days post-Day 1, no biofeedback, just monitoring to test longer-term retention.
  Interventions: Behavioral: Ambulatory voice biofeedback
- Summary feedback (Experimental): Some patients will be assigned (via block randomization) to receive ambulatory voice biofeedback (summary - no cueing, statistics shown every 2 minutes of voicing). Voice monitoring will be conducted for 3 days (device automatically turns off after 42 minutes of voicing): Day 1: biofeedback will be active all day , Day 2: the day after Day 1, no biofeedback, just monitoring to test short-term retention. Day 3: 7 days post-Day 1, no biofeedback, just monitoring to test longer-term retention.
  Interventions: Behavioral: Ambulatory voice biofeedback

INTERVENTIONS:
Behavioral: Ambulatory voice biofeedback — Subjects will be provided cues regarding their vocal behavior in daily life. The cues will either be: 100% feedback = a vibrotactile cue on a smartwatch every time the patient voices incorrectly... 25% feedback = a vibrotactile cue on a smartwatch every 4th time the patient voices incorrectly... Summary feedback = the patient's overall compliance (percentage of voiced time within desired limits) will be presented via a smartwatch every 2 minutes of voicing.

SUMMARY:
This first study will enroll 3 groups of patients with vocal fold nodules that will receive different schedules of ambulatory voice biofeedback (100% frequency feedback, 25% frequency feedback, summary feedback) to avoid their upper 15th percentile of vocal loudness.

DETAILED DESCRIPTION:
We will conduct this study (based on principles of motor learning) using novel smartphone-based ambulatory voice biofeedback systems aimed at improving the carryover of newly established vocal behaviors into daily life. This first study will determine which of three types of ambulatory feedback results in better learning/retention (100% frequency, 25% frequency, or delayed summary feedback every 2 minutes of voicing) of a new vocal behavior (reduced vocal intensity) in three groups of 15 patients with vocal fold nodules. Hypothesis: Patients receiving lower frequency or summary feedback will produce lower initial performance but higher short- and long-term retention than patients receiving feedback 100% of the time.

ELIGIBILITY:
Inclusion Criteria:

Patients with vocal fold nodules

Exclusion Criteria:

Non-English speakers are excluded because prompts on the smartphone app are only available in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Hillman, PhD, Principal Investigator — Mass General Hospital, Harvard, MGH IHP
Locations (1):
- Massachusetts General Hospital - Center for Laryngeal Surgery and Voice Rehabilitation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 100% Frequency | 25% Frequency | Summary Feedback
Started | 10 | 10 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100% Frequency | 25% Frequency | Summary Feedback | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (13) | 24 (8) | 25 (10) | 25 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 29
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 10 | 8 | 7 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 6 | 9 | 6 | 21
  More than one race | 2 | 0 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 9 | 29
Percentage of voicing below threshold [Mean (Standard Deviation); unit: Percentage of voicing below threshold] | 85 (5.97) | 85 (3.21) | 84.75 (5.81) | 84.92 (4.89)

OUTCOME MEASURES:

1. Primary Outcome: Percent Compliance
Description: Percentage compliance is the amount of voiced time patients spent below their biofeedback threshold divided by the total amount of voiced time. Each patient's biofeedback threshold was individually established as their 85th percentile of vocal intensity. Patients were asked to avoid loud voicing, i.e., anything at their 85th percentile or higher. During biofeedback, patients were cued every time (100% frequency) or every 4th time (25% frequency) the voiced louder than their 85th percentile; or provided summary information (their percentage compliance) after every 2 minutes of voicing (summary feedback). During short-term retention monitoring, patients were asked to not voice loud (over or equal to 85th percentile) the next day and the biofeedback was turned off. During long-term retention monitoring, patients were asked to not voice loud one week later without biofeedback.
Time Frame: 1 week
Population: There is a discrepancy in the numbers of enrolled patients here (total = 13) and in previous sections (total = 31). This is because the first 18 patients data were used to refine and adapt study protocols. The final 13 patients data were acquired with this final protocol and we are reporting those data.
Measure: Mean (Standard Deviation); unit: Percentage of voicing below a threshold
Arm/Group | 100% Frequency | 25% Frequency | Summary Feedback
Number analyzed (Participants) | 4 | 5 | 4
Percentage of voicing below a threshold
  Biofeedback | 97.38 (3.72) | 95.11 (3.00) | 94.44 (2.46)
  Short-term Retention | 96.08 (2.26) | 88.86 (10.14) | 90.48 (5.53)
  Long-term Retention | 90.76 (9.29) | 88.39 (7.43) | 90.25 (4.89)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: This is a low-risk clinical trial, as determined by the IRB. We will collect data only on Other Adverse Events, specifically patient-reported skin irritation where the monitor's sensor was taped to the neck during wear. Specifically, each patient will be systematically assessed for skin irritation by the investigator asking the patient if any skin irritation occurred at the end of the study.
Arm/Group | 100% Frequency | 25% Frequency | Summary Feedback
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT03416829/Prot_SAP_000.pdf